CLINICAL TRIAL: NCT01471262
Title: Right and Extended Right Hepatectomy in Patients Beyond 70 Years of Age - Liver Function and Outcome
Brief Title: Right Hepatectomy in Patients Beyond 70 Years Old
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Dr. Emmanuel Melloul, Medical Doctor, Centre Hospitalier Universitaire Vaudois
Other Study IDs: CHV080501
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Complications; Liver Failure, Acute
Keywords: Complications; Mortality; Liver; Failure
MeSH Terms: conditions — Liver Failure, Acute

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Elderly: Patients more or equal to 70 years old
  Interventions: Procedure: Right hepatectomy; Procedure: Extended right hepatectomy
- Young: Patients less than 70 years old
  Interventions: Procedure: Right hepatectomy; Procedure: Extended right hepatectomy

INTERVENTIONS:
Procedure: Right hepatectomy — Right liver resection
  Other Names: Liver surgery
Procedure: Extended right hepatectomy — Right hepatectomy involving 5 or more segments
  Other Names: Liver surgery

SUMMARY:
As a consequence of the increase in life expectancy, hepato-biliary surgeons have to deal with an emerging aged population, which has a potential higher risk for complication and worse long-term outcome. The investigators will be analyzing the liver function and outcome after right or extended right hepatectomy in patients over 70 years old.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Elective right hepatectomy
* Elective extended right hepatectomy

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Other type of hepatectomy
* Emergency hepatectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that will undergo right or extended right hepatectomy for benign or malignant diseases.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2006-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Morbidity | 90 days
  Any type of complication defined according to the Clavien-Dindo Classification of surgical complications.

SECONDARY OUTCOMES:
Mortality | 90 days
  Patient death occuring 90 days post-operatively
Liver failure | 90 days
  Defined according to the Belghiti 50-50 criteria for liver failure.
Hospital stay | 90 days
  Total hospital stay (including re-admission hospital stay) in days

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Melloul, MD, Principal Investigator — Department of Visceral Surgery, University Hospital CHUV, Lausanne, Switzerland; Nicolas Demartines, MD, Study Chair — Department of Visceral Surgery, University Hospital CHUV, Lausanne, Switzerland
Locations (1):
- Department of Visceral Surgery, University Hospital CHUV, Lausanne, Switzerland

REFERENCES:
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Paugam-Burtz C, Janny S, Delefosse D, Dahmani S, Dondero F, Mantz J, Belghiti J. Prospective validation of the "fifty-fifty" criteria as an early and accurate predictor of death after liver resection in intensive care unit patients. Ann Surg. 2009 Jan;249(1):124-8. doi: 10.1097/SLA.0b013e31819279cd. PMID 19106687